CLINICAL TRIAL: NCT04909697
Title: Efficacy of Sivelestat Sodium in the Treatment of ARDS With SIRS, a Multicenter Double-blind Randomized Controlled Clinical Trial
Brief Title: Treatment of ARDS With Sivelestat Sodium
Acronym: TOAWSS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, He Hongli, Principal Investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SichuanPPHospital
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Sham Comparator)
  Interventions: Drug: Saline
- Sivelestat Sodium (Experimental)
  Interventions: Drug: Sivelestat sodium

INTERVENTIONS:
Drug: Sivelestat sodium — 4.8mg/kg sivelestat sodium was given in 50ml normal saline, and was continuously pumped in the dark for 24h, equivalent to 0.2mg/kg/h.Applied for 5 consecutive days
  Arms: Sivelestat Sodium
Drug: Saline — 50ml normal saline was continuously pumped in the dark for 24h. Applied for 5 consecutive days
  Arms: Saline

SUMMARY:
Neutrophil elastase (NE) released by neutrophils play an important role in inflammatory cascade and lung tissue injury of ARDS.Inhibition of NE is expected to prevent the pathophysiological process of ARDS and alleviate lung injury. Siverestat sodium is a specific inhibitor of NE, which has been proved by basic and observational clinical studies to be effective in alleviating lung injury of ARDS, but there is a lack of prospective multi-center randomized controlled clinical trials.Therefore, this study was intended to evaluate the efficacy of sivelestat sodium in the treatment of ARDS patients with SIRS in a multicenter randomized controlled clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Males and females > 18 years old and <75 years old (non-pregnant, non-lactating females).
2. Patients fulfilled the Berlin diagnostic criteria of acute respiratory distress syndrome, with a arterial oxygen partial pressure (PaO2) to fraction of inspired oxygen (FiO2) between 150 mmHg and 300 mmHg.
3. Signed written informed consent has been obtained

Exclusion Criteria:

1. History of chronic respiratory disease
2. Single cardiogenic pulmonary edema
3. Apach2 score ≥21 points
4. Complicated with end-stage disease, or poor prognosis judged by the clinical doctor in charge
5. ARDS course>3 days
6. Agranulocytosis or receiving immunosuppressive agents or high doses of corticosteroids (methylprednisolone>40mg/day)
7. Pregnancy or breastfeeding
8. Participated in this study
9. Do not agree to participate in this experiment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
oxygenation improvement rate | day 3
ventilator free days | day 28

SECONDARY OUTCOMES:
Invasive mechanical ventilation rate | day 28
length of stay in ICU | day 28
length of stay in hospital | day 28
28 days mortality | day 28
ICU mortality | day 28
Incidence of acquired infections | day 28
oxygenation improvement rate | day 1
oxygenation improvement rate | day 5
incidence of severe adverse effect | day 28
activity of neutrophil elastase in plasma | day0
activity of neutrophil elastase in plasma | day 1
activity of neutrophil elastase in plasma | day 3
activity of neutrophil elastase in plasma | day 5
concentration of IL-6 | day 0
concentration of IL-6 | day 1
concentration of IL-6 | day 3
concentration of IL-6 | day 5
concentration of IL-10 | day 0
concentration of IL-10 | day 1
concentration of IL-10 | day 3
concentration of IL-10 | day 5

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Huang, MD, Principal Investigator — Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan provincial people's hospital, Chengdu, Sichuan Privince, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentifed individual participant data are available after the article is published. Data can be accessed with the approval of the authors. Request for data can be made to the corresponding author (drhuangxb@163.com and panchun1982@gmail.com) and will be discussed during a meeting including investigators from all paticipating centers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentifed individual participant data are available after the article is published.
Access Criteria: Data can be accessed with the approval of the authors. Request for data can be made to the corresponding author (drhuangxb@163.com and panchun1982@gmail.com) and will be discussed during a meeting including investigators from all paticipating centers